CLINICAL TRIAL: NCT02895295
Title: Evaluating a Patient-Centered Tool to Help Medicare Beneficiaries Choose Prescription Drug Plans
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Palo Alto Medical Foundation (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, M. Kate Bundorf, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-38241; CDR-1306-03598 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute); 2016.107EXP (Other: Sutter Health Institutional Review Board)
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Prescription Drug Insurance Decision Making
Keywords: Medicare Part D; decision support; prescription drugs; expert recommendation; health insurance choice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Study subjects randomized to the control arm will receive information on how to download their prescription drug information from their electronic medical record and will be provided with a list of resources available in the community to help them choose a prescription drug plan.
  Interventions: Behavioral: Usual Care
- Expert Recommendation (Experimental): Participants randomized to the "Expert Recommendation" arm will receive access to a decision support tool that provides personalized expert scores for particular plans based on individual's likely annual out-of-pocket spending, including plan premiums and spending on prescription drugs, and the Medicare star ratings (a measure of customer satisfaction).
  Interventions: Behavioral: Expert Recommendation
- Individual Analysis (Active Comparator): Participants randomized to "Individual Analysis" arm will receive access to a decision support tool that provides individualized cost information for each plan but not the expert scores for particular plans.
  Interventions: Behavioral: Individual Analysis

INTERVENTIONS:
Behavioral: Expert Recommendation — Decision support tool that provides personalized information on the financial implications of enrolling in different plans and expert recommendations of particular plans.
  Arms: Expert Recommendation
Behavioral: Individual Analysis — Decision support tool that provides personalized information on the financial implications of enrolling in different plans.
  Arms: Individual Analysis
Behavioral: Usual Care — Study subjects randomized to the control arm will receive information on how to download their prescription drug information from their electronic medical record and provided with a list of resources available in the community to help them choose a prescription drug plan.
  Arms: Control

SUMMARY:
The objective of this study is to determine whether providing Medicare beneficiaries with a web-based patient-centered decision tool to help them choose among prescription medication coverage plans improves outcomes for patients including a greater likelihood of changing a plan, better coverage for prescribed drugs, less decisional conflict when choosing plans, and greater satisfaction with the choice process relative to current practice.

DETAILED DESCRIPTION:
In this study, the investigators tested the effectiveness of two versions of a web-based tool (called CHOICE) to help people choose among Medicare Part D plans (Treatments A and B) relative to standard care (Control). Both treatment arms incorporated simplified design and automated importation of an individual's prescription drugs relative to standard care. The treatment arms varied based on whether they provided expert guidance on recommended plans. In the control arm, study participants were directed to the existing, publicly available Medicare.gov website and received instructions on how to download their drugs from the Palo Alto Medical Foundation (PAMF) patient-facing online personal health portal (myhealthonline). The study sample included PAMF patients who were enrolled in Part D plans (not Medicare Advantage) during the 2016 enrollment period. Prior to the 2017 open enrollment period (October 15 to December 7, 2016), we invited a subset of PAMF patients not covered by either MediCal or a Medicare Advantage plan, aged 66-85, residing in 4 counties served by PAMF, and with at least one active medication order to participate in a study examining the effectiveness of decision tools that provide personalized information on the financial implications of enrolling in different Part D plans. The primary study outcomes included 1) Plan switching, 2) Decisional conflict 3) Satisfaction with the choice process, and 4) Change in generosity of coverage of prescription drugs. The investigators measured the primary study outcomes using a combination of administrative data and a post open enrollment survey. The investigators also collected information on individual characteristics at the time of enrollment in the study and implemented a survey examining use of the intervention tool to assess patient experience at the time of use.

ELIGIBILITY:
Inclusion Criteria:

* The study population included Medicare beneficiaries who received care from the Palo Alto Medical Foundation, a large multi-specialty group in the San Francisco Bay Area ages 66-85, one per household enrolled in a Medicare Part D plan in 2016.

Exclusion Criteria:

* Enrolled in a Medicare Advantage Plan and/or MediCal

Ages: 66 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1185 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

REFERENCES:
- [Background] Linder SK, Swank PR, Vernon SW, Mullen PD, Morgan RO, Volk RJ. Validity of a low literacy version of the Decisional Conflict Scale. Patient Educ Couns. 2011 Dec;85(3):521-4. doi: 10.1016/j.pec.2010.12.012. Epub 2011 Feb 5. PMID 21300518

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Study subjects randomized to the control arm will receive information on how to download their prescription drug information from their electronic medical record and provided with a list of resources available in the community to help them choose a prescription drug plan.
  Usual Care: Study subjects randomized to the control arm will receive information on how to download their prescription drug information from their electronic medical record and provided with a list of resources available in the community to help them choose a prescription drug plan.
- Individual Analysis: Participants randomized to "Individual Analysis" arm will receive will receive access to a decision support tool that provides individualized cost information for each plan but not the expert scores for particular plans.
  Individual Analysis: Decision support tool that provides personalized information on the financial implications of enrolling in different plans.
Period: Overall Study
Arm/Group | Control | Expert Recommendation | Individual Analysis
Started | 384 | 410 | 391
Completed | 313 | 316 | 299
Not Completed | 71 | 94 | 92
Not completed — Survey Non-response | 71 | 94 | 92

BASELINE CHARACTERISTICS:
Population: The baseline population represent the number of study participants who completed the final survey administered after the open enrollment period ended.
Groups:
- Control: Usual Care: Study subjects randomized to the control arm received access to information on resources available in the community to help them choose a prescription drug plan and on how to download their prescription drug information from their electronic medical record.
- Expert Recommendation: Study subjects randomized to the "Expert Recommendation" arm received access to a decision support tool that provided personalized, expert recommendations of particular plans as well as personalized information on the financial implications of enrolling in different plans, including plan premiums and spending on prescription drugs, and the Medicare star ratings (a measure of average customer satisfaction).
- Individual Analysis: Study subjects randomized to the "Individual Analysis" arm received access to a decision support tool that provided personalized information on the financial implications of enrolling in different plans, including plan premiums and spending on prescription drugs, and the Medicare star ratings (a measure of average customer satisfaction).
- Total: Total of all reporting groups
Arm/Group | Control | Expert Recommendation | Individual Analysis | Total
Number analyzed (Participants) | 313 | 316 | 299 | 928
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.68 (4.64) | 72.03 (4.55) | 72.11 (4.50) | 72.68 (4.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 150 | 150 | 466
  Male | 147 | 166 | 149 | 462
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 243 | 262 | 240 | 745
  Asian | 35 | 17 | 18 | 70
  Hispanic | 7 | 3 | 6 | 16
  Black | 0 | 1 | 1 | 2
  Other or missing | 28 | 33 | 34 | 95
Estimated prescription drug spending [Mean (Standard Deviation); unit: US dollars] — Estimated spending on prescription drugs for the study respondent given their initial drug list and the features of their 2016 plan including both out-of-pocket spending on prescription drugs and the plan premium. Population: Two survey respondents did not identify their 2016 plan.
  US dollars
    number analyzed (Participants) | 312 | 315 | 299 | 926
    (all) | 1496.80 (1689.97) | 1701.38 (2068.86) | 1580.56 (1493.58) | 1593.44 (1771.73)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Whose 2017 Plan Differed From Their 2016 Plan
Description: Indicator of whether the self-reported plan of the participant differed before and after open enrollment and the participant reported that s/he changed plans during open enrollment.
Time Frame: within 50 days of the end of the open enrollment period.
Population: Set of participants who responded to questions about plan enrollment in the final survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Expert Recommendation | Individual Analysis
Number analyzed (Participants) | 301 | 305 | 290
Participants | 85 | 110 | 86

2. Primary Outcome: Decisional Conflict
Description: Low literacy decisional conflict scale (Linder et al., 2011), edited slightly for context of health insurance rather than treatment choice. The scale has 4 subscales (uncertainty, informed, values clarity and support) with 2 to 3 questions per subscale. Respondents can indicate "yes", "no", or "unsure" for each item. An answer of "yes" receives 0, "unsure" receives 2 and "no" receives 4 points. The sum of the responses to each question within a subscale is normalized to a scale of 25. The subscales are then summed to a total score ranging from 0 to 100 where 0 represents the lowest level of decisional conflict and 100 represents the highest level of decisional conflict.
Time Frame: within 50 days of the end of the open enrollment period.
Population: Study participants who responded to decisional conflict questions on the final survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expert Recommendation | Individual Analysis
Number analyzed (Participants) | 302 | 296 | 285
units on a scale | 21.06 (22.56) | 20.86 (21.99) | 19.56 (22.14)

3. Primary Outcome: Satisfaction With the Choice Process
Description: Response to the question of, "How satisfied are you with the process of choosing a plan?" with 4 potential responses: very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied. The count of participants who responded "very satisfied" is reported.
Time Frame: within 50 days of the end of the open enrollment period
Population: Study participants who responded to question about satisfaction with the choice process on the final survey
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Expert Recommendation | Individual Analysis
Number analyzed (Participants) | 313 | 316 | 299
Participants | 122 | 148 | 134

4. Primary Outcome: Change in Estimated Prescription Drug Spending
Description: Change in estimated prescription drug spending is the difference in estimated spending in US dollars, including both premiums and out-of-pocket spending on prescription drugs, between the participant's 2016 and 2017 plans based on their initial drug list.
Time Frame: within 50 days of the end of the open enrollment period
Population: Study participants who responded to questions about their 2017 plan choice in the final survey administered after open enrollment had ended.
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Control | Expert Recommendation | Individual Analysis
Number analyzed (Participants) | 301 | 305 | 290
US dollars | -178.90 (1029.93) | -249.59 (899.81) | -197.29 (599.38)

ADVERSE EVENTS:
Time Frame: Data were not collected for adverse events or all-cause mortality in this study.
Description: Data were not collected for adverse events or all-cause mortality in this study.
Arm/Group | Control | Expert Recommendation | Individual Analysis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT02895295/Prot_SAP_000.pdf